CLINICAL TRIAL: NCT04124926
Title: A Phase 3, Randomized, Double-Blind, Two Phase, Multicenter Study to Evaluate the Efficacy and Safety of Vonoprazan 20 mg Compared to Lansoprazole 30 mg for Healing in Patients With Erosive Esophagitis and to Evaluate the Efficacy and Safety of Vonoprazan (10 mg and 20 mg) Compared to Lansoprazole 15 mg for the Maintenance of Healing in Patients With Healed Erosive Esophagitis
Brief Title: Efficacy and Safety of Vonoprazan Compared to Lansoprazole in Participants With Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EE-301; 2019-002579-33 (EudraCT Number)
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Results first posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Erosive Esophagitis
Keywords: Erosive Esophagitis; Vonoprazan; Lansoprazole
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Healing Phase: Vonoprazan 20 mg (Experimental): Participants will receive oral vonoprazan 20 mg once per day (QD) for a maximum of 8 weeks.
  Interventions: Drug: Vonoprazan
- Healing Phase: Lansoprazole 30 mg (Active Comparator): Participants will receive oral lansoprazole 30 mg once per day (QD) for a maximum of 8 weeks.
  Interventions: Drug: Lansoprazole
- Maintenance Phase: Vonoprazan 10 mg (Experimental): Participants will receive oral vonoprazan 10 mg once per day (QD) for a maximum of 24 weeks.
  Interventions: Drug: Vonoprazan
- Maintenance Phase: Vonoprazan 20 mg (Experimental): Participants will receive oral vonoprazan 20 mg once per day (QD) for a maximum of 24 weeks.
  Interventions: Drug: Vonoprazan
- Maintenance Phase: Lansoprazole 15 mg (Active Comparator): Participants will receive oral lansoprazole 15 mg once per day (QD) for a maximum of 24 weeks.
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Vonoprazan — Over-encapsulated tablet administered orally with approximately 240 mL water, 30 minutes prior to the morning meal.
  Arms: Healing Phase: Vonoprazan 20 mg; Maintenance Phase: Vonoprazan 10 mg; Maintenance Phase: Vonoprazan 20 mg
Drug: Lansoprazole — Over-encapsulated capsule administered orally with approximately 240 mL water, 30 minutes prior to the morning meal.
  Arms: Healing Phase: Lansoprazole 30 mg; Maintenance Phase: Lansoprazole 15 mg

SUMMARY:
To evaluate the efficacy and safety of vonoprazan compared to lansoprazole in participants with erosive esophagitis.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is ≥18 years of age at the time of informed consent signing.
2. In the opinion of the investigator or subinvestigators, the participant is capable of understanding and complying with protocol requirements.
3. The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures. The participant is informed of the full nature and purpose of the study, including possible risks and side-effects. The participant has the ability to cooperate with the investigator. Ample time and opportunity should be given to read and understand verbal and/or written instructions.
4. The participant is found to have endoscopically confirmed EE of LA Classification Grades A to D during the Screening Period (Visit 1) as assessed by a central adjudicator. The target number of participants with LA classification Grade C or D will be approximately 30% of the total number of participants (300 total). Enrollment of EE participants with Grade A or B will end when the number of participants with Grade A or B EE is approximately 700 or 70% of the total planned number of participants. Given the invasive nature of an endoscopy, any endoscopic confirmation performed in a routine clinical setting before signing the informed consent will be acceptable to use for the purpose of fulfilling the screening requirement if all of the following apply: (1) appropriate endoscopy pictures were taken; (2) appropriate gastric biopsy samples were taken; (3) the endoscopy pictures can be sent to the central adjudicator via the adjudication systems; and (4) all screening procedures (including the completion of adjudication) AND randomization can be completed within a 7-day period after the date of the endoscopy.
5. A female participant of childbearing potential who is or may be sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from the signing of informed consent until 4 weeks after the last dose of study drug.

Exclusion Criteria:

1. The participant's endoscopic examination for entering this study fails to confirm EE within 7 days (no later than 10 days on rare occasion with sponsor approval) prior to randomization.
2. The participant is determined to be positive for Helicobacter pylori (HP) or has had an HP infection within 45 days of randomization.
3. The participant has endoscopic Barrett's esophagus (>1 cm of columnar-lined esophagus) and/or definite dysplastic changes in the esophagus.
4. The participant has any other condition affecting the esophagus, including eosinophilic esophagitis; esophageal varices; viral or fungal infection; esophageal stricture; a history of radiation therapy, radiofrequency ablation, endoscopic mucosal resection, or cryotherapy to the esophagus; or any history of caustic or physiochemical trauma (including sclerotherapy or esophageal variceal band ligation). However, participants diagnosed with Schatzki's ring (mucosal tissue ring around lower esophageal sphincter) are eligible to participate.
5. The participant has scleroderma (systemic sclerosis).
6. The participant has a history of surgery or endoscopic treatment affecting gastroesophageal reflux, including fundoplication and dilation for esophageal stricture (except Schatzki's ring) or a history of gastric or duodenal surgery (except endoscopic removal of benign polyps).
7. The participant has an active gastric or duodenal ulcer at the start of the Screening Period. Additionally, participants with gastric or duodenal erosions are permitted to participate.
8. The participant has received any investigational compound (including those in post marketing studies) within 30 days prior to the start of the Screening Period. A participant who has been screen failed from another clinical study and who has not been dosed may be considered for enrollment in this study.
9. The participant is a study site employee, an immediate family member, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or who may have consented under duress.
10. The participant has cutaneous lupus erythematosus or systemic lupus erythematosus.
11. The participant has had clinically significant upper or lower gastrointestinal bleeding within 4 weeks prior to randomization.
12. The participant has Zollinger-Ellison syndrome or other gastric acid hypersecretory conditions.
13. The participant has a history of hypersensitivity or allergies to vonoprazan (including the formulation excipients: D-mannitol, microcrystalline cellulose, hydroxypropyl cellulose, fumaric acid, croscarmellose sodium, magnesium stearate, hypromellose, macrogol 8000, titanium oxide, or red or yellow ferric oxide), PPIs, or any excipients used in the 13C-urea breath test: mannitol, citric acid, or aspartame. Skin testing may be performed according to local standard practice to confirm hypersensitivity.
14. The participant has a history of alcohol abuse, illegal drug use, or drug addiction within the 12 months prior to screening, or regularly consumes >21 units of alcohol (1 unit = 12 oz/300 mL beer, 1.5 oz/25 mL hard liquor/spirits, or 5 oz/100 mL wine) per week based on self-report. Participants must have a negative urine drug screen at screening.
15. The participant is taking any excluded medications or treatments.
16. If female, the participant is pregnant, lactating, or intending to become pregnant before, during, or within 4 weeks after participating in this study; or intending to donate ova during such time period.
17. The participant has a history or clinical manifestations of significant central nervous system, cardiovascular, pulmonary, hepatic, renal, metabolic, other gastrointestinal, urological, endocrine, or hematological disease that, in the opinion of the investigator, would confound the study results or compromise participant safety.
18. The participant requires hospitalization or has surgery scheduled during the course of the study or has undergone major surgical procedures within 30 days prior to the Screening Visit.
19. The participant has a history of malignancy (including MALToma) or has been treated for malignancy within 5 years prior to the start of the Screening Period (Visit 1). (The participant may be included in the study if he/she has cured cutaneous basal cell carcinoma or cervical carcinoma in situ).
20. The participant has acquired immunodeficiency syndrome or human immunodeficiency virus infection, or tests positive for the hepatitis B surface antigen, hepatitis C virus (HCV) antibody, or HCV RNA. However, participants who test positive for HCV antibody but negative for HCV RNA are permitted to participate.
21. The participant has any of the following abnormal laboratory test values at the start of the Screening Period:

    1. Creatinine levels: >2 mg/dL (>177 μmol/L)
    2. Alanine aminotransferase or aspartate aminotransferase >2 × the upper limit of normal (ULN) or total bilirubin >2 × ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1027 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Phathom Pharmaceuticals
Locations (157):
- United States (109):
  - Pinnacle Research Group, Anniston, Alabama
  - North Alabama Research Center LLC, Athens, Alabama
  - Synexus Clinical Research US, Inc., Birmingham, Alabama
  - Medical Affiliated Research Center Inc, Huntsville, Alabama
  - Synexus Clinical Research US, Inc. - East Valley Family Physicians, PLC, Chandler, Arizona
  - Synexus Clinical Research US, Inc. - Central Arizona Medical Associates, PC, Mesa, Arizona
  - Synexus Clinical Research US, Inc. - Desert Clinical Research, LLC, Mesa, Arizona
  - Elite Clinical Studies - Phoenix - BTC - PPDS, Phoenix, Arizona
  - Hope Research Institute LLC, Phoenix, Arizona
  - Del Sol Research Management - BTC - PPDS, Tucson, Arizona
  - Preferred Research Partners - ClinEdge - PPDS, Little Rock, Arkansas
  - Applied Research Center of Little Rock, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Atria Clinical Research - BTC - PPDS, North Little Rock, Arkansas
  - Anaheim Clinical Trials LLC, Anaheim, California
  - GW Research, Inc. - ClinEdge - PPDS, Chula Vista, California
  - eStudySite - Chula Vista - PPDS, Chula Vista, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - HB Clinical Trials, Inc., Fountain Valley, California
  - OM Research LLC, Lancaster, California
  - Torrance Clinical Research Institute, Lomita, California
  - LA County + USC Medical Center, Los Angeles, California
  - Southern California Research Institute Medical Group, Inc., Los Angeles, California
  - Facey Medical Foundation, Mission Hills, California
  - Palmtree Clinical Research, Palm Springs, California
  - Precision Research Institute, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Paragon Rx Clinical, Inc., Santa Ana, California
  - Synexus Clinical Research US, Inc. - Colorado Springs Family Practice, Colorado Springs, Colorado
  - Western States Clinical Research, Inc., Wheat Ridge, Colorado
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Riverside Clinical Research, Edgewater, Florida
  - Research Centers of America - ERG, Hollywood, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - ENCORE Borland-Groover Clinical Research - ERN - PPDS, Jacksonville, Florida
  - Columbus Clinical Services LLC, Miami, Florida
  - Jesscan Medical Research, Miami, Florida
  - Nuren Medical and Research Center, Miami, Florida
  - Premier Research Associate, Inc., Miami, Florida
  - Gutierrez Medical Center, Orlando, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Synexus Clinical Research US, Inc. - St. Petersburg, Pinellas Park, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Guardian Angel Research Center, Tampa, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Nexgen Research Center, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - In-Quest Medical Research, LLC, Peachtree Corners, Georgia
  - Illinois Gastroenterology Group, Gurnee, Illinois
  - Summit Digestive & Liver Disease Specialists State Street Clinic, Oakbrook Terrace, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Gastroenterology Health Partners, PLLC, New Albany, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - Clinical Trials Management LLC, Covington, Louisiana
  - CroNOLA, LLC., Houma, Louisiana
  - Clinical Trials Management LLC, Metairie, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Meridian Clinical Research, Rockville, Maryland
  - Clinical Associates Research, Towson, Maryland
  - Oakland Medical Research Center, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, PLC, Wyoming, Michigan
  - The Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Heartland Clinical Research, Inc, Omaha, Nebraska
  - Synexus Clinical Research US, Inc. Site 1, Henderson, Nevada
  - Synexus Clinical Research US, Inc. Site 2, Henderson, Nevada
  - Sierra Clinical Research - ClinEdge - PPDS, Las Vegas, Nevada
  - Site 2, Las Vegas, Nevada
  - Las Vegas - Site 1, Las Vegas, Nevada
  - Advanced Research Institute, Reno, Nevada
  - Drug Trials America - ClinEdge, Hartsdale, New York
  - Southtowns Gastroenterology, PLLC, Orchard Park, New York
  - Carolinas Research Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Medication Management LLC, Greensboro, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Peters Medical Research, LLC - ClinEdge - PPDS, High Point, North Carolina
  - Carolina's GI Research, LLC, Raleigh, North Carolina
  - Dayton Gastroenterology, Inc, Dayton, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Rapid City Medical Center LLP, Rapid City, South Dakota
  - Multi Specialty Clinical Research, Johnson City, Tennessee
  - Clinical Research Associates Inc, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Inquest Clinical Research, Baytown, Texas
  - Synexus Clinical Research US, Inc. - Dallas, Dallas, Texas
  - Texas Tech University Health Sciences Center El Paso, El Paso, Texas
  - Precision Research Institute, LLC, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Rio Grande Gastroenterology, McAllen, Texas
  - Digestive System Healthcare, Pasadena, Texas
  - Pearland Physicians, Pearland, Texas
  - Synexus Clinical Research US, Inc., Plano, Texas
  - Quality Research Inc, San Antonio, Texas
  - Gastroenterology Research of San Antonio (GERSA), San Antonio, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Synexus Clinical Research US, Inc., Layton, Utah
  - Advanced Research Institute, Ogden, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - Verity Research, Inc., Fairfax, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Washington Gastroenterology, Bellevue, Washington
  - Harborview Medical Center, University of Washington Medical Center, Seattle, Washington
- Bulgaria (8):
  - Fourth Multiprofile Hospital for Active Treatment, Sofia, Sofia-Grad
  - Multiprofile Hospital for Active Treatment Puls AD - PPDS, Blagoevgrad
  - University Multiprofile Hospital for Active Treatment, Pleven
  - Second Multiprofile Hospital for Active Treatment Sofia, Sofia
  - Medical Center Excelsior OOD - PPDS, Sofia
  - Diagnostic-Consultative Center Aleksandrovska EOOD, Sofia
  - Synexus - Medical Center Synexus Sofia EOOD, Sofia
  - Synexus - Medical Centre Synexus Sofia EOOD, Stara Zagora
- Czechia (5):
  - Nemocnice Pardubickeho kraje, a.s. Orlickoustecka nemocnice, Interni oddeleni, Cs., Ústí nad Orlicí, Pardubice
  - MEDIC KRAL s.r.o., Prague, Prague
  - PreventaMed s.r.o., Olomouc
  - Synexus Czech s.r.o., Prague
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o.z. Oddeleni gastroenterolgie, Ústí nad Labem
- Hungary (7):
  - Debreceni Egyetem Klinikai Kozpont Nagyerdei Krt. 98, Belgyogyaszati Klinika, Debrecen, Hajdú-Bihar
  - Synexus Affiliate BKS Research Kft. Hatvan, Hatvan, Heves County
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Synexus (DRS) - Synexus Magyarország Kft. Budapest, Budapest
  - Synexus Affiliate - Synexus Magyarorszag Kft. Debrecen, Debrecen
  - Synexus (DRS) - Synexus Magyarorszag Kft. Gyula, Gyula
  - Synexus (DRS) - Synexus Magyarország Kft. Zalaegerszeg, Zalaegerszeg
- Poland (19):
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy Centrum Endoskopii Zabiegowej - Poradnia Chorob Jelitowych, Bydgoszcz
  - Gabinet Lekarski-Janusz Rudzinski ul. Powstancow Warszawy 5, Bydgoszcz
  - Synexus - Czestochowa, Częstochowa
  - Synexus - Gdansk, Gdansk
  - Synexus - Gdynia, Gdynia
  - Synexus - Katowice, Katowice
  - Synexus Affiliate - Krakowskie Centrum Medyczne, Krakow
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Sp. J., Ksawerów
  - Synexus - Lodz, Lodz
  - Santa Familia Centrum Badań Profilaktyki i Leczenia, Lodz
  - GASTRO MED Zaklad Opieki Zdrowotnej, Lublin
  - Synexus - Poznan, Poznan
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Twoja Przychodnia - Szczecińskie Centrum Medyczne, Szczecin
  - Gastromed Specjalistyczne Centrum Gastrologii i Endoskopii, Torun
  - REUMATIKA - Centrum Reumatologii NZOZ, Warsaw
  - Synexus - Warszawa, Warsaw
  - Synexus - Wroclaw, Wroclaw
  - Melita Medical, Wroclaw
- United Kingdom (9):
  - Synexus Thames Valley Clinical Research Centre, Reading, Berkshire
  - Synexus - Midlands Clinical Research Centre, Edgbaston, West Midlands
  - Synexus - Wales Clinical Research Centre, Cardiff
  - Synexus - Lancashire Clinical Research Centre, Chorley
  - CPS Research, Glasgow
  - Synexus - Hexham Clinical Research Centre, Hexham
  - Synexus - Merseyside Clinical Research Centre, Liverpool
  - Synexus - Manchester Clinical Research Centre, Manchester
  - Synexus - North Tees Clinical Research Centre, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: Undecided
Data from this study will be published; however, it is undecided if patient level data will be made available at this time.

REFERENCES:
- [Derived] Laine L, DeVault K, Katz P, Mitev S, Lowe J, Hunt B, Spechler S. Vonoprazan Versus Lansoprazole for Healing and Maintenance of Healing of Erosive Esophagitis: A Randomized Trial. Gastroenterology. 2023 Jan;164(1):61-71. doi: 10.1053/j.gastro.2022.09.041. Epub 2022 Oct 10. PMID 36228734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed at 111 sites in 6 countries (Bulgaria, Czechia, Hungary, Poland, the United Kingdom and the United States) between 28 October 2019 and 24 August 2021. Of the 4,167 participants screened for the study, 1,027 participants with erosive esophagitis (EE) were randomized in the Healing Phase.
Pre-assignment Details: Participants were randomized to receive vonoprazan 20 mg once per day (QD) or lansoprazole 30 mg QD using a 1:1 ratio in the Healing Phase. Participants with endoscopic healing of EE at 2 or 8 weeks were re-randomized to receive vonoprazan 10 mg QD, vonoprazan 20 mg QD, or lansoprazole 15 mg QD using a 1:1:1 ratio in the Maintenance Phase.
Groups:
- Healing Phase: Vonoprazan 20 mg: Participants received oral vonoprazan 20 mg QD for a maximum of 8 weeks in the Healing Phase.
- Healing Phase: Lansoprazole 30 mg: Participants received oral lansoprazole 30 mg QD for a maximum of 8 weeks in the Healing Phase.
- Maintenance Phase: Vonoprazan 10 mg: Participants received oral vonoprazan 10 mg QD for 24 weeks.
- Maintenance Phase: Vonoprazan 20 mg: Participants received oral vonoprazan 20 mg QD for 24 weeks.
- Maintenance Phase: Lansoprazole 15 mg: Participants received oral lansoprazole 15 mg QD for 24 weeks.
Period: Healing Phase
Arm/Group | Healing Phase: Vonoprazan 20 mg | Healing Phase: Lansoprazole 30 mg | Maintenance Phase: Vonoprazan 10 mg | Maintenance Phase: Vonoprazan 20 mg | Maintenance Phase: Lansoprazole 15 mg
Started | 514 | 513 | 0 | 0 | 0
Treated With Study Drug | 514 | 510 | 0 | 0 | 0
Completed | 483 | 481 | 0 | 0 | 0
Not Completed | 31 | 32 | 0 | 0 | 0
Not completed — Pretreatment Event, Adverse Event (AE), or Serious AE (SAE) | 3 | 7 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 4 | 0 | 0 | 0
Not completed — Voluntary Withdrawal | 10 | 7 | 0 | 0 | 0
Not completed — Withdrawal of Consent | 5 | 3 | 0 | 0 | 0
Not completed — Miscellaneous | 8 | 7 | 0 | 0 | 0
Not completed — Randomized but not Treated | 0 | 3 | 0 | 0 | 0
Period: Maintenance Phase
Arm/Group | Healing Phase: Vonoprazan 20 mg | Healing Phase: Lansoprazole 30 mg | Maintenance Phase: Vonoprazan 10 mg | Maintenance Phase: Vonoprazan 20 mg | Maintenance Phase: Lansoprazole 15 mg
Started (Re-randomized.) | 0 | 0 | 298 | 298 | 297
Treated With Study Drug | 0 | 0 | 296 | 296 | 297
Completed | 0 | 0 | 274 | 269 | 269
Not Completed | 0 | 0 | 24 | 29 | 28
Not completed — Pretreatment Event, AE, or SAE | 0 | 0 | 3 | 5 | 4
Not completed — Protocol Violation | 0 | 0 | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 7 | 8 | 9
Not completed — Voluntary Withdrawal | 0 | 0 | 3 | 6 | 5
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal of Consent | 0 | 0 | 5 | 5 | 5
Not completed — Miscellaneous | 0 | 0 | 1 | 2 | 4
Not completed — Randomized but not Treated | 0 | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Randomized Set included all participants randomly assigned to receive study drug regardless of whether or not they received a dose of study drug.
Groups:
- Healing Phase: Vonoprazan 20 mg: Participants received oral vonoprazan 20 mg QD for a maximum of 8 weeks in the Healing Phase. Participants were re-randomized to receive vonoprazan 10 mg QD, vonoprazan 20 mg QD, or lansoprazole 15 mg QD using a 1:1:1 allocation ratio in the Maintenance Phase.
- Healing Phase: Lansoprazole 30 mg: Participants received oral lansoprazole 30 mg QD for a maximum of 8 weeks in the Healing Phase. Participants were re-randomized to receive vonoprazan 10 mg QD, vonoprazan 20 mg QD, or lansoprazole 15 mg QD using a 1:1:1 allocation ratio in the Maintenance Phase.
- Total: Total of all reporting groups
Arm/Group | Healing Phase: Vonoprazan 20 mg | Healing Phase: Lansoprazole 30 mg | Total
Number analyzed (Participants) | 514 | 513 | 1027
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 421 | 406 | 827
  >=65 years | 93 | 107 | 200
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 256 | 289 | 545
  Male | 258 | 224 | 482
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 59 | 121
  Not Hispanic or Latino | 450 | 451 | 901
  Unknown or Not Reported | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 474 | 458 | 932
  Black or African-American | 23 | 41 | 64
  Asian | 7 | 6 | 13
  American Indian or Alaska Native | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Other | 5 | 5 | 10
  Unknown | 1 | 1 | 2
  Not Reported | 1 | 0 | 1
Adjudicated Los Angeles (LA) Classification of Esophagitis Grading Scale [Count of Participants; unit: Participants] — LA Classification of Esophagitis Grading Scale:
  * Grade A: One or more mucosal breaks with a length of no longer than 5 mm that did not extend between the tops of 2 mucosal folds.
  * Grade B: One or more mucosal breaks with a length of longer than 5 mm that did not extend between the tops of 2 mucosal folds.
  * Grade C: One or more mucosal breaks that are continuous between the tops of 2 or more mucosal folds, which involves less than 75% of the circumference.
  * Grade D: One or more mucosal breaks, which involves at least 75% of the circumference.
  Participants
    Grade A or B | 337 | 336 | 673
    Grade C or D | 177 | 174 | 351
    Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Healing Phase: Percentage of Participants Who Had Complete Healing of EE by Week 8
Description: A participant was considered to have complete healing of EE if healing was demonstrated during endoscopy.
Time Frame: Week 8
Population: The Modified Intent-to-Treat (MITT) Set (Healing Phase) included all participants randomized into the Healing Phase who had documented EE at baseline and received at least 1 dose of study drug during the Healing Phase. All analyses using the MITT Set grouped subjects according to the randomized treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Healing Phase: Vonoprazan 20 mg | Healing Phase: Lansoprazole 30 mg
Number analyzed (Participants) | 514 | 510
percentage of participants | 92.9 | 84.6
Statistical Analysis 1: Comparison: Healing Phase: Vonoprazan 20 mg vs Healing Phase: Lansoprazole 30 mg; Test type: Non-Inferiority — The noninferiority of vonoprazan to lansoprazole was evaluated with a Farrington and Manning test with a noninferiority margin of 10 percentage points for the difference in EE rates between treatments (vonoprazan minus lansoprazole); p < 0.0001, Farrington and Manning test — 2-sided p-value; difference in percentage = 8.3, 95% CI 2-sided [4.49 to 12.23] — The 2-sided 95% confidence interval (CI) of the difference in EE healing rates between vonoprazan 20 mg and lansoprazole 30 mg was calculated via the Miettinen and Nurminen method

2. Primary Outcome: Maintenance Phase: Percentage of Participants Who Maintained Complete Healing of EE at Week 24
Description: A participant was considered to have complete healing of EE if healing was demonstrated during endoscopy.
Time Frame: Week 24
Population: The MITT Set (Maintenance Phase) included all participants randomized into the Maintenance Phase who had healed EE at the end of the Healing Phase and received at least 1 dose of study drug during the Maintenance Phase. All analyses using the MITT Set grouped participants according to the randomized treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance Phase: Vonoprazan 10 mg | Maintenance Phase: Vonoprazan 20 mg | Maintenance Phase: Lansoprazole 15 mg
Number analyzed (Participants) | 293 | 291 | 294
percentage of participants | 79.2 | 80.7 | 72.0
Statistical Analysis 1: Comparison: Maintenance Phase: Vonoprazan 20 mg vs Maintenance Phase: Lansoprazole 15 mg; Test type: Non-Inferiority — The noninferiority of each dose group of vonoprazan to lansoprazole was evaluated with a Farrington and Manning test with a noninferiority margin of 10 percentage points for the difference in maintenance of healing rates between treatments (vonoprazan minus lansoprazole); p < 0.0001, Farrington and Manning test — 2-sided p-value; difference in percentage = 8.7, 95% CI 2-sided [1.80 to 15.53] — The 2-sided 95% CI of the difference in EE maintenance rates between each vonoprazan group and lansoprazole group was calculated via the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Maintenance Phase: Vonoprazan 10 mg vs Maintenance Phase: Lansoprazole 15 mg; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Farrington and Manning test — 2-sided p-value; difference in percentage = 7.2, 95% CI 2-sided [0.21 to 14.09] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Maintenance Phase: Vonoprazan 20 mg vs Maintenance Phase: Lansoprazole 15 mg; Test type: Superiority — The superiority of the vonoprazan 20 mg group to lansoprazole group p-value was evaluated with a Farrington and Manning test with the null hypothesis difference ≤0 versus the alternative hypothesis difference >0; p = 0.0136, Farrington and Manning test — 2-sided p-value
Statistical Analysis 4: Comparison: Maintenance Phase: Vonoprazan 10 mg vs Maintenance Phase: Lansoprazole 15 mg; Test type: Superiority — The superiority of the vonoprazan 10 mg group to lansoprazole group p-value was evaluated with a Farrington and Manning test with the null hypothesis difference ≤0 versus the alternative hypothesis difference >0; p = 0.0436, Farrington and Manning test — 2-sided p-value

3. Secondary Outcome: Healing Phase: Percentage of 24-hour Heartburn-free Days
Description: A 24-hour heartburn-free day was defined as a day having no heartburn among all diary entries for that day. The percentage of 24-hour heartburn-free days was calculated using all days with at least 1 evening or morning diary entry during the treatment period of this phase.
Time Frame: Day 1 to Week 8
Population: The MITT Set (Healing Phase) including only participants with at least one heartburn diary entry.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Healing Phase: Vonoprazan 20 mg | Healing Phase: Lansoprazole 30 mg
Number analyzed (Participants) | 509 | 507
percentage of days | 66.8 (34.60) | 64.1 (35.46)
Statistical Analysis 1: Comparison: Healing Phase: Vonoprazan 20 mg vs Healing Phase: Lansoprazole 30 mg; Test type: Non-Inferiority — If the lower bound of the CI was greater than -15%, noninferiority would be concluded; difference in mean percentage = 2.7, 95% CI 2-sided [-1.60 to 7.03] — The 2-sided 95% CI of the difference in mean percentage of 24-hour heartburn-free days between vonoprazan 20 mg and lansoprazole 30 mg was calculated from Welch's t-test

4. Secondary Outcome: Healing Phase: Percentage of Participants With Baseline LA Classification Grades C or D Who Had Complete Healing of EE at Week 2
Description: A participant was considered to have complete healing of EE if healing was demonstrated during endoscopy.
  LA Classification of Esophagitis Grading Scale:
  Grade C: One or more mucosal breaks that are continuous between the tops of 2 or more mucosal folds, which involves less than 75% of the circumference.
  Grade D: One or more mucosal breaks, which involves at least 75% of the circumference.
Time Frame: Week 2
Population: The MITT Set (Healing Phase) including only participants with baseline LA Classification Grades C or D.
Measure: Number; unit: percentage of participants
Arm/Group | Healing Phase: Vonoprazan 20 mg | Healing Phase: Lansoprazole 30 mg
Number analyzed (Participants) | 177 | 174
percentage of participants | 70.2 | 52.6
Statistical Analysis 1: Comparison: Healing Phase: Vonoprazan 20 mg vs Healing Phase: Lansoprazole 30 mg; Test type: Superiority — [test comment as in outcome 2, analysis 3]; p = 0.0008, Farrington and Manning test — 2-sided p-value; difference in percentage = 17.6, 95% CI 2-sided [7.44 to 27.43] — The 2-sided 95% CI of the difference in EE healing rates between vonoprazan 20 mg and lansoprazole 30 mg was calculated via the Miettinen and Nurminen method

5. Secondary Outcome: Healing Phase: Percentage of Participants With Onset of Sustained Resolution of Heartburn by Day 3
Description: Sustained resolution was defined as at least 7 consecutive days with no daytime or night time heartburn as assessed by the daily diary. A participant was considered to have sustained resolution of heartburn by Day 3 if the first day of the 7 consecutive days without symptoms was on Days 1, 2, or 3.
Time Frame: Day 1 to maximum of Day 10 (inclusive of 7 day heartburn assessment)
Population: The MITT Set (Healing Phase) included all participants randomized into the Healing Phase who had documented EE at baseline and received at least 1 dose of study drug during the Healing Phase. All analyses using the MITT Set grouped subjects according to the randomized treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Healing Phase: Vonoprazan 20 mg | Healing Phase: Lansoprazole 30 mg
Number analyzed (Participants) | 514 | 510
percentage of participants | 34.4 | 32.2
Statistical Analysis 1: Comparison: Healing Phase: Vonoprazan 20 mg vs Healing Phase: Lansoprazole 30 mg; Test type: Superiority — [test comment as in outcome 2, analysis 3]; p = 0.4392, Farrington and Manning test — 2-sided p-value; difference in percentage = 2.3, 95% CI 2-sided [-3.50 to 8.04] — The 2-sided 95% CI of the difference in sustained resolution rates between vonoprazan 20 mg and lansoprazole 30 mg was calculated via the Miettinen and Nurminen method

6. Secondary Outcome: Healing Phase: Percentage of Participants With Baseline LA Classification Grades C or D Who Had Complete Healing of EE by Week 8
Description: as for outcome 4
Time Frame: Week 8
Population: The MITT Set (Healing Phase) including only participants with baseline LA Classification Grades C or D.
Measure: Number; unit: percentage of participants
Arm/Group | Healing Phase: Vonoprazan 20 mg | Healing Phase: Lansoprazole 30 mg
Number analyzed (Participants) | 177 | 174
percentage of participants | 91.7 | 72.0
Statistical Analysis 1: Comparison: Healing Phase: Vonoprazan 20 mg vs Healing Phase: Lansoprazole 30 mg; Test type: Superiority — Observed p-value and not a formal test per the preplanned fixed-sequence testing procedure. The superiority of the vonoprazan 20 mg group to lansoprazole group p-value was evaluated with a Farrington and Manning test with the null hypothesis difference ≤0 versus the alternative hypothesis difference >0; p < 0.0001, Farrington and Manning test — 2-sided p-value; difference in percentage = 19.6, 95% CI 2-sided [11.84 to 27.58] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Healing Phase: Percentage of Participants Who Had Complete Healing of EE at Week 2
Description: A participant was considered to have complete healing of EE if healing was demonstrated during endoscopy.
Time Frame: Week 2
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Healing Phase: Vonoprazan 20 mg | Healing Phase: Lansoprazole 30 mg
Number analyzed (Participants) | 514 | 510
percentage of participants | 74.3 | 68.2
Statistical Analysis 1: Comparison: Healing Phase: Vonoprazan 20 mg vs Healing Phase: Lansoprazole 30 mg; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.0348, Farrington and Manning test — 2-sided p-value; difference in percentage = 6.1, 95% CI 2-sided [0.53 to 11.60] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: Maintenance Phase: Percentage of Participants With Baseline LA Classification Grades C or D Who Maintained Complete Healing of EE at Week 24
Description: as for outcome 4
Time Frame: Week 24
Population: The MITT Set (Maintenance Phase) including only participants with baseline LA Classification Grades C or D with nonmissing data.
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance Phase: Vonoprazan 10 mg | Maintenance Phase: Vonoprazan 20 mg | Maintenance Phase: Lansoprazole 15 mg
Number analyzed (Participants) | 95 | 92 | 96
percentage of participants | 74.7 | 77.2 | 61.5
Statistical Analysis 1: Comparison: Maintenance Phase: Vonoprazan 20 mg vs Maintenance Phase: Lansoprazole 15 mg; Test type: Superiority — [test comment as in outcome 2, analysis 3]; p = 0.0196, Farrington and Manning test — 2-sided p-value; difference in percentage = 15.7, 95% CI 2-sided [2.50 to 28.44] — The 2-sided 95% CI of the difference in maintenance rates between each vonoprazan group and lansoprazole 15 mg group was calculated via the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Maintenance Phase: Vonoprazan 10 mg vs Maintenance Phase: Lansoprazole 15 mg; Test type: Superiority — [test comment as in outcome 2, analysis 4]; p = 0.0490, Farrington and Manning test — 2-sided p-value; difference in percentage = 13.3, 95% CI 2-sided [0.02 to 26.14] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Maintenance Phase: Percentage of 24-hour Heartburn-free Days
Description: as for outcome 3
Time Frame: Day 1 to Week 24
Population: The MITT Set (Maintenance Phase) including only participants with at least one heartburn diary entry.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Maintenance Phase: Vonoprazan 10 mg | Maintenance Phase: Vonoprazan 20 mg | Maintenance Phase: Lansoprazole 15 mg
Number analyzed (Participants) | 291 | 290 | 294
percentage of days | 80.9 (28.59) | 80.6 (29.96) | 78.6 (27.49)
Statistical Analysis 1: Comparison: Maintenance Phase: Vonoprazan 20 mg vs Maintenance Phase: Lansoprazole 15 mg; Test type: Non-Inferiority — If the lower bound of the CI was greater than -15%, noninferiority would be concluded; difference in mean percentage = 2.0, 95% CI 2-sided [-2.63 to 6.72] — The 2-sided 95% CI of the difference in mean percentage of 24-hour heartburn-free days between each vonoprazan group and the lansoprazole group was calculated from Welch's t-test
Statistical Analysis 2: Comparison: Maintenance Phase: Vonoprazan 10 mg vs Maintenance Phase: Lansoprazole 15 mg; Test type: Non-Inferiority — If the lower bound of the CI was greater than -15%, noninferiority would be concluded; difference in mean percentage = 2.3, 95% CI 2-sided [-2.27 to 6.84] — [estimate comment as in outcome 9, analysis 1]

ADVERSE EVENTS:
Time Frame: Healing Phase: Day 1 to Week 8; Maintenance Phase: Day 1 to Week 28
Description: The Safety Set included all randomized participants who received at least 1 dose of study drug. All analyses using the Safety Set grouped subjects according to the treatment actually received.
Arm/Group | Healing Phase: Vonoprazan 20 mg | Healing Phase: Lansoprazole 30 mg | Maintenance Phase: Vonoprazan 10 mg | Maintenance Phase: Vonoprazan 20 mg | Maintenance Phase: Lansoprazole 15 mg
All-Cause Mortality (participants affected / at risk) | 0/514 | 0/510 | 0/296 | 2/296 | 0/297
Serious Adverse Events (participants affected / at risk) | 3/514 | 3/510 | 10/296 | 14/296 | 7/297
Other Adverse Events (participants affected / at risk) | 50/514 | 46/510 | 72/296 | 81/296 | 74/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healing Phase: Vonoprazan 20 mg (N=514) | Healing Phase: Lansoprazole 30 mg (N=510) | Maintenance Phase: Vonoprazan 10 mg (N=296) | Maintenance Phase: Vonoprazan 20 mg (N=296) | Maintenance Phase: Lansoprazole 15 mg (N=297)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatolithiasis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healing Phase: Vonoprazan 20 mg (N=514) | Healing Phase: Lansoprazole 30 mg (N=510) | Maintenance Phase: Vonoprazan 10 mg (N=296) | Maintenance Phase: Vonoprazan 20 mg (N=296) | Maintenance Phase: Lansoprazole 15 mg (N=297)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 13 (13) | 3 (3) | 7 (7) | 13 (14)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 2 (2) | 4 (4) | 10 (12) | 3 (3)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 9 (9) | 4 (4) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 11 (12) | 12 (12) | 8 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 2 (2) | 7 (7) | 11 (12) | 6 (6)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 7 (8)
COVID-19 (Infections and infestations) | 8 (8) | 6 (6) | 12 (12) | 26 (26) | 18 (18)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3) | 7 (7) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6) | 4 (4) | 8 (8) | 1 (1) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 6 (6) | 8 (8) | 4 (4)
Hypertension (Vascular disorders) | 3 (3) | 4 (4) | 9 (9) | 8 (9) | 6 (6)
Headache (Nervous system disorders) | 6 (6) | 6 (6) | 3 (3) | 2 (2) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04124926/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT04124926/SAP_001.pdf